CLINICAL TRIAL: NCT00433368
Title: Efficacy of a Three Days' Infusion of L-Ornithine-L-Aspartate as an Adjuvant Therapy in Cirrhotic Patients With Overt Hepatic Encephalopathy: A Placebo Controlled Study
Brief Title: Efficacy of L-Ornithine-L-Aspartate in Cirrhotics With Hepatic Encephalopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OA001
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Hepatic Encephalopathy
Keywords: L-ornithine-L-aspartate,; porto-systemic encephalopathy,; hepatic encephalopathy,; liver cirrhosis,; mental state
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis | interventions — ornithylaspartate

INTERVENTIONS:
Drug: L-Ornithine L-Aspartate

SUMMARY:
The purpose of this study is to determine whether L-Ornithine L-Aspartate is effective for the improvement of Overt Hepatic Encephalopathy.

DETAILED DESCRIPTION:
There is no effective treatment available for hepatic encephalopathy at the moment; therefore we aimed to check the efficacy and safety of L-ornithine L-aspartate(LOLA). It provides critical substrates for ureagenesis and glutamine synthesis, the two primary mechanisms by which the body rids itself of excess ammonia. Ornithine is a specific activator of ornithine carbamyl transferase and carbamylphosphate synthetase, and, in addition, is a substrate for ureagenesis. These reactions are carried out mainly in the periportal portion of the hepatic lobules. Aspartate and ornithine, after conversion to alfa-ketoglutarate, are substrates for glutamine synthesis, which is performed exclusively by a small population of perivenous hepatocytes, the so-called perivenous scavenger cells. The ammonia lowering effect resulting from the stimulation of these two basic mechanisms of ammonia detoxification has been studied in animals and was confirmed in humans in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis, diagnosed on the basis of clinical findings, sonographic, and/or histologic basis,
* Patients >14 years, with HE grades 1 to 4 according to West Haven Criteria,
* Hyperammonemia (fasting venous blood ammonia level >60 µmol/l), and
* Patients with a single reversible precipitating factor of HE such as constipation, hypokalemia, urinary tract infection, respiratory tract infection, spontaneous bacterial peritonitis (SBP), dehydration, or none.

Exclusion Criteria:

* hepatocellular carcinoma,
* severe septicemia,
* active gastrointestinal bleeding,
* hepatorenal syndrome,
* acute superimposed liver injury,
* advanced cardiac or pulmonary disease and end stage renal failure,
* patients with minimal HE
* patients taking sedatives, antidepressants, or benzodiazepines and
* patients with chronic HE on metronidazole or lactulose prior to admission.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108
Dates: Start 2003-10; Study Completion 2004-09

PRIMARY OUTCOMES:
Improvement in HE grade.
deterioration in HE grade.

SECONDARY OUTCOMES:
Length of hospital stay
fasting ammonia level and
mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Jafri, MD; FRCP, Study Chair — Chairman Department of Medicine, Aga Khan University Hospital; Shahab Abid, MD, Principal Investigator — Associate Professor, Department of Medicine, Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] [1] ] STAEDT U, LEWELING H, GLADISCH R, KORTSIK C, HAGMULLER E, HOLM E. Effects of ornithine aspartate on plasma ammonia and plasma amino acids in patients with cirrhosis. A double-blind, randomized study using a four-fold crossover design. J Hepatol 1993;19(3): 424-430. [2] KIRCHEIS G, NILIUS R, HELD C, BERNDT H, BUCHNER M, GÖRTELMEYER R, et al. Therapeutic efficacy of L-ornithine-L-aspartate infusions in patients with cirrhosis and hepatic encephalopathy: results of a placebo-controlled, double-blind study. Hepatology 1997;25(6):1351-1360. [3] FEHÉR J, LÁNG I, GÓGL A, VARGA L, TOMPOS G, PRÓNAI L. Effect of ornithine-aspartate infusion on elevated serum ammonia concentration in cirrhotic patients - results of a randomized, placebo-controlled double-blind multicentre trial. Med Sci Monit 1997; 3(5):669-673. [4] KIRCHEIS G, WETTSTEIN M, VOM DAHL S, HÄUSSINGER D. Clinical efficacy of L-ornithine-L-aspartate in the management of hepatic encephalopathy. Met Brain Dis 2002;17(4): 453-462. [5] REES CJ, OPPONG K, AL MARDINI H, HUDSON M, RECORD CO. Effect of L- ornithine-L-aspartate on patients with and without TIPS undergoing glutamine challenge: a double blind, placebo controlled trial. Gut 2000; 47(4): 571-574.